CLINICAL TRIAL: NCT05360342
Title: Incorporation of Vitamin K Into Uremic Lipoproteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jürgen Floege, Univ.-Prof. Dr. med., RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RWTH Aachen University
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Vitamin K Deficiency
MeSH Terms: conditions — Vitamin K Deficiency | interventions — Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin K supplement (Experimental): Administration of a single dose vitamin K
  Interventions: Drug: Vitamin K supplement

INTERVENTIONS:
Drug: Vitamin K supplement — Single dose of vitamin K supplement
  Other Names: High dose vitamin K1 and K2 supplement

SUMMARY:
Chronic kidney disease (CKD) patients have an increased cardiovascular risk with corresponding cardiovascular calcifications. CKD patients exhibit a functional vitamin K deficiency. Calcification can be prevented by vitamin K intake. The aim of this study is to investigate the cause for the vitamin K deficiency beyond a diminished dietary vitamin K uptake.

DETAILED DESCRIPTION:
This study is a monocentric, 1-armed interventional trial. Participants will be recruited at the University Hospital of the RWTH Aachen.

We will analyse serially collected serum from 10 dialysis patients, after ingestion of a single vitamin K supplement, compared to healthy controls. Lipoprotein fractions will be isolated and the corresponding vitamin K contents will be measured by chromatography.

The vitamin K supplement contains 3 subforms of vitamin K: vitamin K1 (1000µg), menaquinone-4 (1000µg) and menaquinone-7 (200µg).

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Controls: adequate kidney function (GFR > 60 ml/min/1,73m2)
* Patients: chronic haemodialysis
* Written consent to take part in the study

Exclusion criteria

* Intake of vitamin K antagonists
* gastro-intestinal diseases interfering with vitamin K intake
* profound anemia with an Hb < 10 g/dl
* judicial or official commitment to an institution
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Vitamin K content in lipoproteins | 1 year
  Assessment of vitamin K incorporation into lipoproteins

SECONDARY OUTCOMES:
PIVKA-II levels | 1 year
  PIVKA-II in serum as assessed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Floege, MD, Principal Investigator — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No